CLINICAL TRIAL: NCT03630731
Title: Maintenance Treatment of Chidamide in Chemotherapy-responded Stage IV or Relapsed/Refractory Extranodal Natural Killer/T-cell Lymphoma, Nasal Type
Brief Title: Maintenance Treatment of Chidamide in Stage IV or Relapsed/Refractory Extranodal NK/T-cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mei Dong, Medical doctor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCCRENT
Record Dates: First submitted 2018-08-07; First posted 2018-08-15 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Natural Killer/T-Cell Lymphoma, Nasal and Nasal-Type
MeSH Terms: interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: chidamide — For those who responded to induction chemotherapy, chidamide will be given OR orally 30mg biw for at least half a year

SUMMARY:
Extranodal natural killer/T-cell lymphoma, nasal type (NKTCL) is a highly aggressive peripheral T-cell lymphoma (PTCL). Patients with newly diagnosed stage IV and relapsed/refractory have poor prognosis. 5-year progression-free survival was reported only 55%. Chidamide is a selective histone deacetylase inhibitor which was approved by FDA in treating relapsed or refractory PTCL. In phase I and II studies of chidamide, patients with relapsed or refractory NKTCL achieved a higher overall remission. Patients who obtained complete or partial remission had much favourable duration of remission. Thus, the invesgator design this study to evaluate the role of maintenance treatment of chidamide for induction chemotherapy-responded newly-diagnosed advanced and relapsed/refractory NKTCL patients.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of NKTCL with typical morphology and immunophenotype, according to the 2008 World Health Organization classification of lymphomas;
2. newly-diagnosed stage IV disease or relapsed or refractory disease；
3. age ≥ 18 years;
4. ECOG performance status 0-2;
5. at least one measurable lesion;
6. adequate hematological, hepatic, and renal functions; e.g., absolute neutrophil count ≥ 1.5 × 109/L, platelet count ≥ 80 × 109/L, total bilirubin ≤ 1.5 × upper limit of normal, alanine transaminase and aspartate transaminase ≤ 2 × upper limit of normal, and creatinine ≤ 1.5 mg/dl;
7. life expectancy of more than 3 months.

Exclusion Criteria:

1. Patients with newly-diagnosed stage I-II disease;
2. pregnancy or lactation;
3. any coexisting medical problems of sufficient severity to prevent full compliance with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
PFS | 1 year
  PFS was defined as the period from the date of treatment till the date of disease progression, relapse, or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Mei Dong, Principal Investigator — Cancer Hospital Chinese Academy of Medical Science
Locations (1):
- Cancer Hospital and Institute, Chinese Academy of Medical Sciences (CAMS) and Peking Union Medical College (PUMC), Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes